CLINICAL TRIAL: NCT01595464
Title: A Randomized Controlled Study of Mind-Body Skills Groups for the Treatment of War-Related Trauma in Adults in Gaza
Brief Title: Mind-Body Skills Groups for the Treatment of War-Related Trauma in Adults in Gaza
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Center for Mind-Body Medicine (Other)
Collaborators: The Atlantic Philanthropies (Other)
Responsible Party: Principal Investigator, James S. Gordon, M.D., Founder and Director, The Center for Mind-Body Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GA-CMBM-001
Record Dates: First submitted 2012-05-08; First posted 2012-05-10 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mind-Body Skills Groups (Experimental)
  Interventions: Behavioral: Mind-Body Skills Groups
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Mind-Body Skills Groups — Teaching mind-body skills such as meditation, biofeedback, guided imagery, and meditation in a group setting
  Arms: Mind-Body Skills Groups

SUMMARY:
The objective of this study is to determine whether participation in a mind-body skills program by war-traumatized adults in Gaza will result in improvement of posttraumatic stress symptoms and depression, and will increase posttraumatic growth compared to a control group.

ELIGIBILITY:
Inclusion Criteria:

* having experienced a political violence or war-related criterion A stressor
* meeting the American Psychiatric Association (DSM-IV TR) criteria for PTSD according to screening scores on the PTSD Checklist- Civilian version

Exclusion Criteria:

* former psychosocial or medical treatment for mental health conditions
* significant cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2012-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
PTSD Checklist-Civilian Version | Change from Baseline (Week 1) at 11 weeks
PTSD Checklist-Civilian Version | Change from Week 11 at 23 weeks
PTSD Checklist-Civilian Version | Change from Baseline (Week1) at 23 Weeks

SECONDARY OUTCOMES:
Center for Epidemiological Studies Depression Scale (CES-D) | Change from Baseline (Week 1) at 11 weeks
Center for Epidemiological Studies Depression Scale (CES-D) | Change from Week 11 at 23 weeks
Center for Epidemiological Studies Depression Scale (CES-D) | Change from Baseline (Week1) at 23 Weeks
Posttraumatic Growth Inventory | Change from Baseline (Week 1) at 11 weeks
Posttraumatic Growth Inventory | Change from Week 11 at 23 weeks
Posttraumatic Growth Inventory | Change from Baseline (Week1) at 23 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: James S Gordon, MD, Principal Investigator — The Center for Mind-Body Medicine
Locations (1):
- The Center for Mind-Body Medicine, Gaza City, Palestine, Israel

REFERENCES:
- See also: The Center for Mind-Body Medicine website — http://www.cmbm.org